CLINICAL TRIAL: NCT02734030
Title: Knee Extensor Muscle Inhibition and Neuromechanical and Morphological Properties in Young Women Symptomatic and Asymptomatic for Anterior Knee Pain
Brief Title: Knee Extensor Muscle Properties in Young Women Symptomatic and Asymptomatic for Anterior Knee Pain
Status: Completed | Type: Observational
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Marco Aurélio Vaz, PhD, PhD, Federal University of Rio Grande do Sul
Other Study IDs: UFRGS - 1.032.452
Record Dates: First submitted 2016-01-26; First posted 2016-04-12 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Anterior Knee Pain Syndrome
Keywords: Anterior Knee Pain Syndrome; Quadriceps Femoris; Muscle Inhibition; Interpolated Twitch Technique; Muscle Architecture; Single Leg Squat; Women Knee Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Group: Knee pain-free females with no history of lower limb injuries serving as a control group.
  .
- Anterior Knee Pain Group: Females with anterior knee pain syndrome were enrolled in this group.

SUMMARY:
This study aims to compare the knee extensors' mechanical, morphological and myoelectric properties between subjects affected by anterior knee pain and a healthy control group. The investigators hypothesis is that patients with anterior knee pain present a reduction in the knee extensors' mechanical, morphological and myoelectric properties due to chronic muscle inhibition produced by the syndrome. In addition, the study also aims to evaluate whether there are differences in methodology for application of the Interpolated Twitch Technique for evaluation of the quadriceps muscle inhibition by comparing the use of supramaximal electrical stimulation on the femoral nerve (gold standard) with stimulation on the motor point (new methodology) in healthy subjects and individuals affected by anterior knee pain. The investigators hypothesis is that the stimulation on the motor point is less discomfortable than on the femoral nerve and muscle inhibition results are less variable (with lower dispersion) due to such lower discomfort

DETAILED DESCRIPTION:
Participants were divided in two groups (control group, n=16 and anterior knee pain group, n=16). Prior to participation, informed consent was obtained from all subjects. The evaluation was performed at the lower limb with severe symptoms of anterior knee pain in the patients, and at the dominant limb in the control group. Quadriceps Muscle inhibition was estimated using the Interpolated Twitch Technique, which involves applying a single electrical twitch stimulation to the femoral nerve (gold standard) during a maximal isometric knee extensor contraction. Muscle inhibition measurements were obtained with the aid of a Grass S88 (Quincy, MA, USA.) Muscle Stimulator in combination with and isolation unit approved for human use. Isometric and isokinetic knee extensor torques were obtained with a Biodex System 3 dynamometer (Biodex Medical System, Shirley - NY, USA). Electromyographic muscle activity was measured with bipolar surface electrodes (Kendall, Meditrace - 100; Ag/AgCl) that were placed on the muscle bellies of vastus medialis, vastus lateralis and rectus femoris. Muscle architecture was measured with a B-mode ultrasonographic system (SSD; Aloka Inc., Tokyo, Japan) with a linear-array probe (60 mm, 7.5MHz; Aloka). Single Leg Squat was used for clinical evaluation of the lower limb functionality.

ELIGIBILITY:
Inclusion Criteria:

* Anterior Knee pain group:

  1. Retropatellar or peripatellar knee pain in at least 2 of the following functional activities: stair ascent or descent, running, kneeling, squatting, prolonged sitting, jumping;
  2. Score smaller than 85 points on the Kujala Questionnaire;
  3. Physically active according to the International Physical Activity Questionnaire (IPAQ - short version)
  4. Body mass index less than 30
* Control group:

  1. Knee pain-free females with no history of lower limb injuries

Exclusion Criteria:

1. Body mass index higher than 30
2. Sedentary subjects
3. Cardiovascular, neurological or cognitive disorders
4. Any cardiorespiratory, neuromuscular, or metabolic disease that could represent an absolute contraindication or a contraindication to the performance of maximum strength tests
5. Previous surgery on lower limb
6. Participation in a strength-training programme or physiotherapy treatment for knee injuries in the past six months
7. Otherwise associated injury in the lower limb joints other than anterior knee pain syndrome
8. Pregnancy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young women symptomatic and assymptomatic for anterior knee pain syndrome
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Torque | Torque was measured during a single visit to the laboratory during the study.The evaluation was performed up to 5 months
  Torque is an expression of the muscular strength and was assessed by dynamometry.
Muscular architecture | Muscle architecture was measured one time during the study. The evaluation was performed up to 5 months
  Muscular architecture (muscle thickness, pennation angle and fascicle length) was assessed by ultrasonography
Muscle inhibition | Muscle inhibition was measured during a single visit to the laboratory during the study. The evaluation was performed up to 5 months
  Quadriceps muscle inhibition was assessed using the Interpolated Twitch Technique comparing the use of supramaximal electrical stimulation on the femoral nerve (gold standard) with stimulation on the motor point (new methodology).
Muscular electrical activation | Muscular electrical activation was measured during a single visit to the laboratory during the study. The evaluation was performed up to 5 months
  Electrical activation was assessed by surface electromyography (EMG)
Patellofemoral cartilage thickness | Patellofemoral cartilage thickness was measured one time during the study. The evaluation was performed up to 5 months
  Patellofemoral cartilage thickness were assessed by ultrasonography
Single Leg Squat | Single leg squat performance was measured one time during the study. The evaluation was performed up to 5 months
  Single leg squat was measured with a video camera and allowed to determine lower limb functionality

SECONDARY OUTCOMES:
Knee pain | Knee pain during the tests was measured after all knee extensor contractions. The evaluation was performed up to 5 months.
  Knee pain was measured with a Visual Analogue Scale

CONTACTS AND LOCATIONS:
Overall Officials: Marco Vaz, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Exercise Research Laboratory, School of Physical Education, Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No